CLINICAL TRIAL: NCT02798679
Title: Cardiac Fibrosis and Risk Prediction in Cancer Treatment-Related Cardiotoxicity
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: CV-2016-24434
Record Dates: First submitted 2016-05-12; First posted 2016-06-14 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether pre-existing cardiac fibrosis is a predictor of cancer treatment-related cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer or lymphoma with a >2 year life expectancy
* A treatment plan that includes anthracyclines and/or trastuzumab
* Age >45 years
* Able to hold breath for 10 seconds
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Refusal or inability to provide informed consent
* Known heart failure or LVEF <50%
* Heart rate over 100 bpm
* Renal dysfunction with GFR <30 mL/min/1.73m2
* Participants with pacemakers, defibrillators, functioning neurostimulator devices or other implanted electronic devices
* Symptomatic claustrophobia
* Plans to move within 24 months of enrollment

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive participants with breast cancer or lymphoma scheduled to receive anthracycline-based chemotherapy or trastuzumab.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Cardiotoxicity assessed clinically or by cardiac MRI | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Chetan Shenoy, MBBS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No